CLINICAL TRIAL: NCT01098773
Title: Pulmonary and Cardiac Ultrasound During Weaning From Mechanical Ventilation
Acronym: PULCO
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-0069; 2009-A01310-57 (Other: Afssaps)
Record Dates: First submitted 2010-04-01; First posted 2010-04-05 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Adult Patients Ventilated More Than 48 h; Stable Respiratory and Hemodynamic Conditions for SBT; Consent of Patients; Arterial Line
Keywords: Weaning from mechanical ventilation; BNP; Lung ultrasound; Echocardiography

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- patients requiring ventilation
- patients who weaned permanently

SUMMARY:
Prospective observational clinical multicentric study in ICU with ventilated patients requiring chest ultrasound analysis.

DETAILED DESCRIPTION:
Prospective observational clinical multicentric study on ICU ventilated patients requiring chest ultrasound analysis during weaning from mechanical ventilation with 48 hours of follow-up. Studying variations of cardiac markers

ELIGIBILITY:
Inclusion Criteria:

- Adult patients ventilated more than 48 h

* Stable respiratory and hemodynamic conditions for SBT
* Consent of patients
* Arterial line

Exclusion Criteria:

* Laryngeal dyspnea
* Tracheostomy
* Arythmya
* No echogenicity
* Paraplegia >T8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational clinical multicentric study on ICU ventilated patients requiring chest ultrasound analysis during weaning from mechanical ventilation with 48 hours of follow-up. Studying variations of cardiac markers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Compare the change in pulmonary aeration during the test of weaning from mechanical ventilation (before, at the end, and 4-6 h after) between patients requiring re-ventilation before the 48th hour, and those weaned permanently. | before, at the end, and 4-6 h after
  Compare the change in pulmonary aeration during the test of weaning from mechanical ventilation (before, at the end, and 4-6 h after) between patients requiring re-ventilation before the 48th hour, and those weaned permanently.

SECONDARY OUTCOMES:
Studying variations, during weaning from mechanical ventilation, of pressure of left ventricle filling (E / Ea) coupled with those of plasma BNP. | in the 4-6 early hours
  Studying variations, during weaning from mechanical ventilation, of pressure of left ventricle filling (E / Ea) coupled with those of plasma BNP.
Assessing the effects of E / Ea and BNP variations on the success or failure in the 4-6 early hours. | in the 4-6 early hours.
  Assessing the effects of E / Ea and BNP variations on the success or failure in the 4-6 early hours.
Compare the variations of lung ultrasound score during the test of the weaning from mechanical ventilation between patients failed the spontaneous breathing test (SBT) and those extubated after successful SBT. | in the 4-6 early hours
  Compare the variations of lung ultrasound score during the test of the weaning from mechanical ventilation between patients failed the spontaneous breathing test (SBT) and those extubated after successful SBT.
Comparison of levels epithelial and endothelial markers | at h0, h1, h4, h6
Constitution serum bank for epithelial (sRAGE) markers dosages | at h0, h1, h4, h6
constitution serum bank for endothelial (angiopoietin) markers dosages | at h0, h1, h4, h6

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien PERBET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Jabaudon M, Perbet S, Pereira B, Soummer A, Roszyk L, Guerin R, Futier E, Lu Q, Bazin JE, Sapin V, Rouby JJ, Constantin JM. Plasma levels of sRAGE, loss of aeration and weaning failure in ICU patients: a prospective observational multicenter study. PLoS One. 2013 May 27;8(5):e64083. doi: 10.1371/journal.pone.0064083. Print 2013. PMID 23724022